CLINICAL TRIAL: NCT02305472
Title: Clinical Evaluation of a Bioresorbable Sirolimus-eluting Coronary Scaffold in the Treatment of Patients With de Novo Coronary Artery Lesion (NeoVas): a Single Arm Registry Study
Brief Title: NeoVas Bioresorbable Coronary Scaffold Registry Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lepu Medical Technology (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPM-201403
Record Dates: First submitted 2014-11-27; First posted 2014-12-02 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2015-12

CONDITIONS: Coronary Artery Disease
Keywords: NeoVas; Bioresorbable Coronary Scaffold; Sirolimus; Registry Trial
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NeoVas BCS (Experimental): The NeoVas sirolimus-eluting bioresorbable coronary scaffold system is a PLLA-based polymer scaffold and contains the antiproliferative drug sirolimus.
  Interventions: Device: NeoVas BCS

INTERVENTIONS:
Device: NeoVas BCS — Subjects receiving NeoVas BCS
  Other Names: NeoVas Bioresorbable Coronary Scaffold

SUMMARY:
The NeoVas Bioresorbable Coronary Scaffold Registry Trial is a prospective, multi-center, single arm registry trial based on the NeoVas FIM study which verified the safety and effectiveness of NeoVas initially. This study is to evaluate the safety and effectiveness of NeoVas sirolimus-eluting bioresorbable coronary scaffold in the treatment of patients with de novo coronary lesion.

DETAILED DESCRIPTION:
Approximately 825 subjects will be enrolled and receive NeoVas BCS(Lepu Medical Technology (Beijing) Co.,Ltd). Subjects will have clinical follow-up at 30, 90, 180 and 270 days and at 1,2,3,4 and 5 years. The primary endpoint is target lesion failure(TLF) at 1 year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age must be 18-75 years, men or unpregnant women.
* Patient must have evidence of myocardial ischemia, suitable for elective PCI. Subjects with stable angina or silent ischemia and <70% diameter stenosis must have objective sign of ischemia as determined by one of the following, echocardiogram, nuclear scan, ambulatory ECG or stress ECG. In the absence of noninvasive ischemia, fractional flow reserve(FFR) must be done and indicative of ischemia.
* Patients with one or two de novo lesions located in different epicardial vessels.
* Target lesion must be≤20mm in length(visual estimation)and 2.75 to 3.75 mm in diameter(Online QCA).
* Target lesion is with a visually estimated stenosis of ≥70%(or≥50% and evidence of myocardial ischemia) with a TIMI flow of ≥1.
* The target lesion can be covered by one scaffold(except the rescue scaffold).
* Patient must be an acceptable candidate for coronary artery bypass graft.
* Patient or a legally authorized representative must provide written Informed Consent prior to any study related procedure.

Exclusion Criteria:

* Patients has had a known diagnosis of acute myocardial infarction(AMI) within 7 days preceding the procedure; CK and CK-MB have not returned within normal limits at the time of procedure.
* Chronic total occlusion lesions (TIMI 0 grade blood flow prior to implantation), left trunk vessel lesion, ostial lesion, multi-branch lesions needing treated, bifurcation lesion (diameter ≥2.0mm, branch opening stenosis exceeds 50% or need balloon expansion) and bridge vessel lesions; there is thrombus visible in the target blood vessels.
* Severe calcified lesions and twisted lesions which cannot be pre-expanded, and lesions unsuitable for delivering and expanding stents.
* In-stent restenosis lesion.
* Patient has undergone previous stenting anywhere within the target vessel(s) within the previous 12 months, or will require stenting within the target vessel(s) within 1 year after the study procedure; target vessels that has been implanted with stents.
* Severe heart failure(over NYHA III grade ), or left ventricular ejection fraction(LVEF)<40%( supersonic inspection or left ventricular radiography ).
* Known renal insufficiency(eGFR<60 ml/min, serum creatinine>2.5mg/dL, or subject on dialysis).
* Patients with hemorrhage tendency, an active digestive ulcer history, a cerebral hemorrhage or subarachnoid hemorrhage history, or cerebral apoplexy within half a year, and these patients who contraindicate against platelet inhibitors and anticoagulant therefore cannot bear anticoagulation treatment.
* Patient has a known hypersensitivity or contraindication to aspirin, clopidogrel, ticagrelor or prasugrel, heparin, contrast agent, polylactic acid or sirolimus that cannot be adequately pre-medicated.
* Life expectancy < 12 months.
* Patient is participating in another device or drug study that has not reached the primary endpoint of the study.
* Patient's inability to fully cooperate with the study protocol.
* Patient has a heart transplant.
* Patient has current unstable arrhythmias, such as high risk ventricular premature beat and ventricular tachycardia.
* Patient is receiving or scheduled to receive chemotherapy for malignancy within 30 days prior to or after the procedure.
* Patient is receiving immunosuppression therapy and has known immunosuppressive or autoimmune disease.
* Patient is receiving or scheduled to receive chronic anticoagulation therapy (e.g., heparin, warfarin).
* Elective surgery is planned within the first 6 months after the procedure that will require discontinuing either aspirin, clopidogrel, ticagrelor or prasugrel.
* Platelet count<100,000 cells/mm3 or>700,000 cells/mm3, a WBC of<3,000 cells/mm3, or documented or suspected liver disease.
* Patient has extensive peripheral vascular disease that precludes safe 6 French sheath insertion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 825 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Target lesion failure | 1 year
  Target lesion failure is a composite endpoint of cardiac death, target vessel related myocardial infarction (TV-MI) and the ischemia-driven target lesion revascularization.

SECONDARY OUTCOMES:
Device Success | intraoperative
  Successful delivery and deployment of the assigned scaffold at the intended target lesion and successful withdrawal of the delivery system with attainment of final in-scaffold residual stenosis of less than 30% by quantitative coronary angiography (QCA) (by visual estimation if QCA unavailable). The success or failure of the first-aid stent is not included.
Procedural Success | At time of procedure up to 7 days in hospital
  Achievement of final in-scaffold residual stenosis of less than 30% by QCA (by visual estimation if QCA unavailable) with successful delivery and deployment of at least one assigned scaffold at the intended target lesion and successful withdrawal of the delivery system for the target lesion without the occurrence of cardiac death, target vessel MI or repeat TLR. For the circumstance of two target lesions, both lesions must meet the success criteria.
Target lesion failure | 30days, 3,6,9 months and 2,3,4,5 years
  Target lesion failure is a composite endpoint of cardiac death, target vessel related myocardial infarction (TV-MI) and the ischemia-driven target lesion revascularization.
Patient oriented composite endpoint | 30days, 3,6,9 months and 1,2,3,4,5 years
  Patients oriented composite endpoint includes all-cause death, all myocardial infarction and any revascularization.
Ischemia-driven Target Lesion Revascularization (iTLR) | 30 days, 3,6,9 months and 1, 2, 3, 4, 5 years
Ischemia-driven Target Vessel Revascularization (iTVR) | 30 days, 3,6,9 months and 1, 2, 3, 4, 5 years
All coronary revascularization (PCI and CABG) | 30 days, 3,6,9 months and 1, 2, 3, 4, 5 years
Scaffold thrombosis | 30 days, 3,6,9 months and 1, 2, 3, 4, 5 years
  Scaffold thrombosis will be categorized as acute (≤1day), subacute (>1day ≤30 days) and late (>30 days).Clinical presentation of acute coronary syndrome with angiographic evidence of scaffold thrombosis (angiographic appearance of thrombus within or adjacent to a previously treated target lesion).In the absence of angiography, any unexplained death, or acute MI (ST segment elevation or new Q-wave) in the distribution of the target lesion within 30 days.
Percentage of patients who experienced angina | 30days, 3,6,9 months and 1, 2, 3, 4, 5 years
  Angina is defined as any angina or angina equivalent symptoms determined by the physician and/or research coordinator after interview of the patient, and as adjudicated by a clinical events committee (CEC).

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, MD, Study Chair — The general hospital of Shenyang military region; Guosheng Fu, Principal Investigator — Sir Run Run Shaw Hospital; Bo Xu, Principal Investigator — Beijing Fuwai hospital, National center for cardiovascular diseases China; Yao-Jun Zhang, Principal Investigator — Nanjing First Hospital, Nanjing Medical University
Locations (27):
- China (27):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - General Hospital of Armed Police Forces, Beijing, Beijing Municipality
  - Aerospace Center Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Nanfang Hospital Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Bethune Peace Hospital of PLA, Shijiazhuang, Hebei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Wuhan General Hospital of Guangzhou Military, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Nanjing Drum Tower Hospital, the Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The general hospital of Shenyang military region, Shenyang, Liaoning
  - Renji Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Tenth People'S Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Changhai Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Xijing Hospital, the Fourth Military Medical University, Xi’an, Shanxi
  - The First Affiliated Hospital of Xi'An Jiaotong University, Xi’an, Shanxi
  - Chengdu Military General Hospital, Chengdu, Sichuan
  - Affiliated Hospital of The Chinese People's Armed Police Forces Logistic College, Tianjin, Tianjin Municipality
  - Tianjin first center hospital, Tianjin, Tianjin Municipality
  - Kunming General Hospital of Chengdu Military Region, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital,School of Medicine, Zhejiang University, Hangzhou, Zhejiang